CLINICAL TRIAL: NCT01065272
Title: Dexamethasone Versus Placebo in the Treatment of Viral Bronchiolitis in Patients With Either Eczema and or Parental or Sibling History of Asthma.A Randomized Controlled Trial.
Brief Title: Dexamethasone in the Treatment of Bronchiolitis in Patients With Either Eczema and or Family History of Asthma
Acronym: #9105
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #9105/09; #9105/09 (Other: Hamad Medical Corporation)
Record Dates: First submitted 2010-01-12; First posted 2010-02-09 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2012-09

CONDITIONS: Bronchiolitis
Keywords: Dexamethasone; Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Dexamethasone; Steroids; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ventolin - Dexamethasone group (Active Comparator): Ventolin nebulization with normal saline is given at 0,30,60,120 and 180 minutes,then every 2 hourly. Oral Dexamethasone is also given daily for 5 days.
  Interventions: Drug: Dexamethasone
- Ventolin - Placebo group (Placebo Comparator): Ventolin nebulization with normal saline is given at 0,30,60,120 and 180 minutes,then every 2 hourly. Oral Placebo is also given daily for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — 0.5 ml Salbutamol in 2 ml normal saline is given at 0,30,60,120,180 minutes and then every 2 hourly till discharge.
  1mg/kg of oral Dexamethasone with cherry flavour is also given in the first day, then 0.6 mg/kg/day for 4 days
  Other Names: Steroids
  Arms: Ventolin - Dexamethasone group
Drug: Placebo — 0.5 ml Salbutamol in 2 ml normal saline is given at 0,30,60,120,180 minutes and then every 2 hourly till discharge.
  1mg/kg of oral Placebo is also given in the first day, then 0.6 mg/kg/day for 4 days
  Other Names: normal saline plus cherry flavour
  Arms: Ventolin - Placebo group

SUMMARY:
The investigators hypothesized that oral Dexamethasone in addition to nebulized Salbutamol will improve the Bronchiolitis Clinical Severity Score,duration of treatment in the short stay unit,need for hospitalization and readmissions to the pediatric emergency in a subgroup of patients diagnosed as Bronchiolitis with either eczema and or a parental or sibling history of Asthma.

Two groups randomized will be given Nebulized Ventolin plus either oral Dexamethasone or placebo for 5 days.

Bronchiolitis severity score plus vital signs will be recorded regularly until patient is fit for discharge.

Patients will be discharged on Ventolin inhaler and to complete the five days course of oral Dexamethasone Patients will be followed up for 7 days post discharge by telephone.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blinded controlled study. It will be conducted in the main Pediatric Emergency Centre in Qatar(Al- Saad),during the period of Jan 2010 - April 2012.

The study has been approval by the Institution Research Board. The sample size will be 200 patients.100 patients in each arm.

Patients triaged as moderate to severe bronchiolitis will be evaluated and eligible patients are admitted to short stay unit and managed as usual. History and full physical examination will be done by the attending physician and the nurse will check 02 sat., respiratory rate and pulse rate.

The Bronchiolitis clinical severity score will be assessed and then guardians of eligible patients will be approached explaining the purpose and treatment modalities.

Patients will be included after obtaining a verbal and written consent. A CXR and an RSV test will be done for all study patients upon recruitment. The attending physician will complete the data collection sheet A computer generated randomization code will be prepared by the statistician. A pharmacist will prepare the study medications and the placebo. Patients will be randomized to either one of the two treatments:- Ventolin-Dexamethasone group: Oral Dexamethasone 1mg/kg will be given for the first day and then 0.6mg/kg for the next 4 days in addition to the Ventolin nebulizations.

Ventolin-Placebo group: Oral Placebo with a volume equivalent to that of Dexamethasone will be given for the first day and then for the next 4 days in addition to the Ventolin nebulizations.

Nebulized Ventolin 0.5ml in 2 ml Normal Saline will also be given at 0, 30, 60, 120 and 180 minutes and then every 2hours.

Bronchiolitis severity score and O2 saturation will be recorded at enrollment, then after 4,6 and 12hours then every 12 hourly until discharged.

To give additional Ventolin nebulization will be decided clinically as per the discretion of the treating physician and will be recorded.

Nebulized epinephrine will not be used except if the patient is severely distressed. Nebulized Epinephrine 0.5 mg/kg (max 5mg/dose) mixed in 3ml normal saline will be allowed for severely distressed patients as an add on therapy given on PRN basis..

Additional interventions such as Oxygen therapy, Intravenous fluids and PRN nebulized Epinephrine will be recorded as additional therapies.

Patients fit for discharge will have their nebulization stopped & date, time documented.

Physician will discharge patients based on clinical grounds as not needing supplemental oxygen,minimal or no chest recessions,minimal wheezing or crackles and feeding adequately Patients will be sent home on Ventolin inhaler 2 puffs q 4 hours for 48 hours Then 2 puffs every 4 hours when needed plus the study medication syrup to complete 5days course.

Follow up for one-week post discharge by a phone call daily will be conducted and patients will be assessed in PEC when needed.

ELIGIBILITY:
Inclusion Criteria:

* Infant's ≥ 4weeks and ≤ 18 month.
* First time wheezers.
* Bronchiolitis clinical severity score ≥ 4.
* History of eczema in the patient.
* Parenteral history of asthma
* Sibling history of asthma

Exclusion Criteria:

* Prematurity (Gestational age 34 weeks or less).
* Previous history of wheezing episode.
* Use of steroids within the last 48 hours.
* Critically ill patients with one or more of the following:

  * Obtunded consciousness,
  * Progressive respiratory failure requiring PICU admission.
  * History of apnea.
  * Oxygen saturation less than 85%.
* Chronic lung disease of prematurity.
* Cystic fibrosis.
* Congenital heart disease.
* Immunodeficiency.
* Exposure to Varicella within 21 days before enrollment.

Ages: 4 Weeks to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Patients diagnosed as bronchiolitis were discharged at 12 hours for each group | 12 hours

SECONDARY OUTCOMES:
Patients diagnosed as bronchiolitis were discharged at 18, 24 , 36 and 48 hours for each group | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Khalid M Al-Ansari, FRCPC,FAAP, Principal Investigator — Hamad Medical Corporation, Weill Cornell Medical College, Doha-Qatar
Locations (1):
- Hamad Medical Corporation, Pediatric Emergency Center,Alsaad., Doha, Baladīyat ad Dawḩah, Qatar